CLINICAL TRIAL: NCT04907305
Title: Next-Gen MS: A Prospective, Cluster-randomized Study Evaluating the Impact of "Feed-forward" Patient Reported Outcomes Data to Clinical Teams Managing Adults Living With MS in a Learning Health System for MS Research
Brief Title: Next-Gen MS: Feed-forward PRO Data for MS Research
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to change in strategic priorities.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Other Study IDs: MS200077_0013
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Multiple Sclerosis; Patient Reported Outcomes; Patient Determined Disease Steps; Learning Healthcare System
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Feed-forward PRO: Participants in this group will participate in monthly learning collaborative webinars. Feed-forward of patient reported outcomes (PRO) data collected from the main study (NCT04735406) will be used.
- Control Group (Usual Care): Participants in the control group will receive usual care practices during the clinical encounters.

SUMMARY:
This Next Generation learning health system for Multiple Sclerosis (Next-Gen MS) study is a sub-study of the MS-LINK™ Outcomes Study (NCT04735406). The study aims to examine the effects of using feed forward Patient Reported Outcomes (PROs) data in real-world Multiple Sclerosis (MS) care settings. The study will be conducted within an emerging Learning Healthcare System (LHS).

ELIGIBILITY:
Inclusion Criteria:

* Participants willing and able to provide written informed consent
* Participants with clinical diagnosis of Multiple Sclerosis (MS)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants from United States with Multiple sclerosis (MS) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1594 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Health-Related Quality of Life 14 Item (HR-QoL-14) | Baseline up to 18 Months

SECONDARY OUTCOMES:
Percentage of Participants with >=1-point Increase from Baseline in Patient Determined Disease Steps (PDDS) Sustained Via Consecutive Measures Over 3 Months | Baseline up to 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (8):
- United States (8):
  - Alabama Neurology Associates, Birmingham, Alabama
  - Georgetown University, Washington D.C., District of Columbia
  - Atlanta Neuroscience Institute, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The Memorial Hospital, d.b.a Memorial Healthcare, Owosso, Michigan
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - The University of Texas of Austin, Austin, Texas
  - The University of Texas Health Science Center, San Antonio, Texas

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200077_0013
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html